CLINICAL TRIAL: NCT02185235
Title: To Evaluate The Efficacy of Electrical Stimulation and Biofeedback Treatment for Pelvic Floor Disorder Women
Brief Title: A Randomized Controlled Trial of Electrical Stimulation to Treat Pelvic Floor Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Principal Investigator, Tsung-Hsien Su, Mackay Memorial Hospital, Mackay Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14MMHIS031
Record Dates: First submitted 2014-06-11; First posted 2014-07-09 (Estimated); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Pelvic Organ Prolapse; Incontinence
Keywords: Electrical stimulation; Biofeedback
MeSH Terms: conditions — Pelvic Organ Prolapse | interventions — Electric Stimulation; Biofeedback, Psychology

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Biofeedback & Electrical Stimulation (Experimental): Twice a week, 20 minutes for each time. One course includes 18 times treatment.
  Interventions: Device: Electrical Stimulation; Device: Biofeedback
- Biofeedback & Pelvic Floor Training (Active Comparator): Pelvic floor training every 20 minutes for each time, twice a week. and total for 18 times.
  Interventions: Device: Biofeedback; Other: Pelvic Floor Training

INTERVENTIONS:
Device: Electrical Stimulation — The Chartered Society of Physiotherapy recommends the following standard for electrical devices.
  Frequency: 35 Hertz. Pulse width: 250µs (0.25ms). Current type: bi-phasic rectangular. Intensity: maximum tolerated. Duty-cycle: 5 seconds on/10 seconds off. Very weak muscles: 5 seconds on/15 seconds off.
  Treatment time: 5 minutes initially, gradually increasing to 20 minutes.
  Other Names: Femiscan Stim (Mega Electronics Ltd)
  Arms: Biofeedback & Electrical Stimulation
Device: Biofeedback — Biofeedback is a treatment technique in which people are trained to improve their health by using signals from their own bodies
  Other Names: Femiscan Multi-trainer
Other: Pelvic Floor Training — First, as you are sitting or lying down, try to contract the muscles you would use to stop urinating To contract the pelvic muscles, squeeze for 3 seconds and then relax for 3 seconds.
  Repeat this exercise to 20 minutes each session.
  Arms: Biofeedback & Pelvic Floor Training

SUMMARY:
Female pelvic floor disorders (PFDs) include urinary incontinence,pelvic organ prolapse (POP), and fecal incontinence-which often occur together.

Pelvic floor disorders impair multiple aspects of the life quality, including the sexual function of women.

Surgery became the first choice of treatment, however, and not until 1980s was the renewed interest in conservative therapies.

This may be because of higher awareness among women and cost of and morbidity after surgery.

The conservative treatment included pelvic floor muscle training, electrical stimulation, vaginal cones, and biofeedback.

The outcome was up to 35~70 % improved rate as the literature before. Current guidelines recommended conservative management as a first-line therapy. However, there was no consistent consensus on this issue due to variations in stimulation parameters、adjuvant concurrent modality or duration of treatment course, and insufficient result about large and long term follow up of randomized- controlled studies.

Therefore, the investigators try to conduct one randomized-controlled trial to evaluate the efficacy of conservative treatment for Pelvic floor disorder (Pelvic organ prolapse, urinary incontinence, chronic pelvic pain etc.).

At the aspect of Quality of life, our studies tried to focus on the different domains of pelvic disorder and sexual quality by means of validated questionnaire more objectively.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from pelvic organ prolapse and/or urinary incontinence and/or fecal incontinence.

Exclusion Criteria:

* Patient is pregnant The patient had any major medical or psychiatric disease The patient with Metabolic medical device

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-06; Primary Completion 2024-06 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
1-Hour Pad test of urine leakage amount (gm) | Total 18 times of treatment, for 3 months
  A pad test is a tool to used to measure urine leakage amount . Pad testing can be done over a period of time to one hour.
  A sanitary napkin is weighed and then worn for sixty minutes, during which time the individual is asked to perform certain activities which may include:
  * Walking briskly for three minutes
  * Sitting and then standing ten to twenty times
  * Walking up and down stairs for one to two minutes
  * Picking up objects from the floor five to ten times
  * Coughing twelve times (at various strengths; may be repeated)
  * Running in place for one minute (may be repeated) The pad is then removed and weighed again to calculate the amount of urine voided.

SECONDARY OUTCOMES:
Quality of life (score) | Total 18 times of treatment, for 3 months

OTHER OUTCOMES:
Vaginal pressure (mmHg) | Total 18 times of treatment, for 3 months
  Use the vaginal probe sensor to evaluate the objective level of vaginal squeezing pressure and endurance time
Urodynamics data analysis | Total 18 times of treatment, for 3 months
  Use urodyanmic examinations for evaluation of bladder function

CONTACTS AND LOCATIONS:
Overall Officials: TSUNG H Su, Professor, Principal Investigator — Mackay Memorial Hospital
Locations (1):
- Taiwan, Taipei, Mackay Memorial hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Lau HH, Lai CY, Hsieh MC, Peng HY, Chou D, Su TH, Lee JJ, Lin TB. Effect of intra-vaginal electric stimulation on bladder compliance in stress urinary incontinence patients: the involvement of autonomic tone. Front Neurosci. 2024 Aug 7;18:1432616. doi: 10.3389/fnins.2024.1432616. eCollection 2024. PMID 39170685